CLINICAL TRIAL: NCT01040299
Title: Combine Mechanized Gait Trainer and Transcranial Direct Current Stimulation in Chronic Stroke Patients: Randomized Control Trial
Brief Title: Mechanized Gait Trainer Combine Transcranial Galvanic Stimulation (tDCS) in Chronic Stroke
Acronym: GT-1-tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT-1-tDCS
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Hemiparesis; Cerebrovascular Disorders
Keywords: GangTrainer; Gait Rehabilitation; Cerebrovascular Disorders; Robot assisted; Transcranial direct current stimulation
MeSH Terms: conditions — Paresis; Cerebrovascular Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GangTrainer and tDCS (Experimental): The experimental group patients receive a total of 10 treatments of repetitive locomotor training with electromechanical gait device (duration 30 min) + tDCS (duration first 7 min) with the anodal electrode is place over the presumed lower limb area of the lesioned hemisphere, and the cathodal electrode is place above the controlateral orbital.
  Interventions: Device: GangTrainer and tDCS
- control group1 (Sham Comparator): The control group 1 receive a total of 10 treatments with only GT (duration 30 min) with sham-stimulation.
  Interventions: Device: control group1
- control group2 (Active Comparator): The control group 2 receive a total of 10 treatments with convectional physiotherapy.
  Interventions: Other: Control group2

INTERVENTIONS:
Device: GangTrainer and tDCS — The experimental group patients receive a total of 10 treatments of repetitive locomotor training with electromechanical gait device (duration 30 min) + tDCS (duration first 7 min) with the anodal electrode is place over the presumed lower limb area of the lesioned hemisphere, and the cathodal electrode is place above the controlateral orbital.
  Arms: GangTrainer and tDCS
Device: control group1 — The control group 1 receive a total of 10 treatments with only GT (duration 30 min) with sham-stimulation.
  Other Names: GangTrainerGT1
  Arms: control group1
Other: Control group2 — The control group 2 receive a total of 10 treatments with convectional physiotherapy.
  Other Names: convectional physiotherapy
  Arms: control group2

SUMMARY:
Transcranial galvanic stimulation (tDCS), seems to promote motor recovery after stroke by stimulating (anodal) or inhibiting (cathodal) neural circuits in the brain. In the treatment of severe lower limb paresis after stroke, the GangTrainer GT1 (GT) proved to be effective, but nevertheless only a few patients could use their affect lower limb functionally in daily life on deambulation after robot training. Therefore the present study intends to combine both approaches, tDCS + GT, apply at the same time every day for two weeks in order to improve the effectiveness of GangTrainer therapy in the gait rehabilitation.

DETAILED DESCRIPTION:
Transcranial galvanic stimulation (tDCS), seems to promote motor recovery after stroke by stimulating (anodal) or inhibiting (cathodal) neural circuits in the brain. In the treatment of severe lower limb paresis after stroke, the GangTrainer GT1 (GT) proved to be effective. Therefore the present study intends to combine both approaches, tDCS + GT, apply at the same time every day for two weeks in order to improve the effectiveness of GangTrainer therapy in the gait rehabilitation. The rehabilitation programme are compose 3 kinds of locomotor training interventions (experimental group, control group 1 and control group 2).

During intervention experimental group, patients receive a total of 10 treatments of repetitive locomotor training with electromechanical gait device (duration 30 min) + tDCS (duration first 7 min) with the anodal electrode is place over the presumed lower limb area of the lesioned hemisphere, and the cathodal electrode is place above the controlateral orbital. The anodal stimulation is expected to facilitate the activity of the lower limb motor area side directly, while the cathodal stimulation of the non-lesioned hemisphere is expected to facilitate the lesioned side indirectly by decreasing inhibitory inputs. The control group 1 receive a total of 10 treatments with only GT (duration 30 min) with sham-stimulation, and the control group 2 receive a total of 10 treatments with convectional physiotherapy

ELIGIBILITY:
Inclusion Criteria:

* European Stroke scale between 75-85
* First time supratentorial, ischaemic or hemorrhagic stroke.
* Diagnosis of ischemic brain injury or intracerebral hemorrhage by MRI or computed tomography > 6 months after the onset of stroke.
* Age < 80 years.
* Ability to stand upright, supported or unsupported, for 1 minute.
* Patients with ischaemic or haemorrhagic stroke.
* In-patient participating in a comprehensive rehabilitation programme.
* patients written informed consent of participation in the study approved by the local ethical committee.
* absence of cardiac, psychological and orthopedic conditions that might interfere with the result.

Exclusion Criteria:

* Preceding epileptic fits.
* an EEG suspect of elevated cortical excitability.
* a sensitive scalp skin.
* severe cognitive impairment.
* metallic implants within the brain.
* previous brain neurosurgery.
* medications altering the level of cortical excitability
* medications with a presumed positive or negative effect on brain plasticity.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Motricity Index | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.

SECONDARY OUTCOMES:
Barthel Index | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
European Stroke Scale | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Modified Ashworth Scale | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Questionary of Ambulation | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Rivermead Motor Assessment Score | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Functional Ambulation Category | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Ten Meters Walking Test | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Six Minutes Walking Test | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Spatia-temporal Gait analysis | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Motricity Index | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania Nicola Smania, Doctor, Principal Investigator
Locations (1):
- Azienta Ospedaliera, SSO Rehabilitation Unit, Verona, Verona, Italy, Verona, Italy

REFERENCES:
- [Background] Hesse S, Werner C, Schonhardt EM, Bardeleben A, Jenrich W, Kirker SG. Combined transcranial direct current stimulation and robot-assisted arm training in subacute stroke patients: a pilot study. Restor Neurol Neurosci. 2007;25(1):9-15. PMID 17473391
- [Result] Pohl M, Werner C, Holzgraefe M, Kroczek G, Mehrholz J, Wingendorf I, Hoolig G, Koch R, Hesse S. Repetitive locomotor training and physiotherapy improve walking and basic activities of daily living after stroke: a single-blind, randomized multicentre trial (DEutsche GAngtrainerStudie, DEGAS). Clin Rehabil. 2007 Jan;21(1):17-27. doi: 10.1177/0269215506071281. PMID 17213237
- [Result] Dias D, Lains J, Pereira A, Nunes R, Caldas J, Amaral C, Pires S, Costa A, Alves P, Moreira M, Garrido N, Loureiro L. Can we improve gait skills in chronic hemiplegics? A randomised control trial with gait trainer. Eura Medicophys. 2007 Dec;43(4):499-504. PMID 18084173